CLINICAL TRIAL: NCT01690208
Title: Evaluation of Morbidities, Endpoints and Reaching Targets in Diabetic Patients Managed by an All-encompassing Program Led by a Diabetes Specialist Team
Brief Title: Evaluation of Morbidities, Endpoints and Reaching Targets in Diabetic Patients Managed by a Diabetes Specialist Team
Acronym: EMERALD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Asia Diabetes Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRE-2012.136-T
Record Dates: First submitted 2012-09-19; First posted 2012-09-21 (Estimated); Last update posted 2015-08-10 (Estimated); Status verified 2015-08

CONDITIONS: Diabetes; Obesity
Keywords: Diabetes; Structure Care
MeSH Terms: conditions — Diabetes Mellitus; Obesity | interventions — fluoro-emerald

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- EMERALD (Experimental): Patients assigned to the EMERALD group will be invited to join the multi-component program which will last for 1 year. This program will be held on a 4-weekly basis for the first 3-4 months followed by a maintenance program involving 2-4 group activities every year. Between clinic visits, patients in this group will also receive telephone reminders from the staff and peer supporters to reinforce compliance and for social support.
  Interventions: Other: EMERALD
- Usual Care (Active Comparator): Irrespective of the assignment group, all patients will undergo a baseline comprehensive assessment using the JADE portal disease management system. All patients will also receive a 2-hour session on how to interpret their individualised JADE report and risk profiles, whilst the importance of achieving targets and optimizing self care will be reinforced.
  Patients assigned to the UC group will be followed up in their usual clinic according to the 'standard' practice.
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: EMERALD — Patients assigned to the EMERALD group will be followed up at a Diabetes Centre led by the nurses and supported by diabetologists, with a particular emphasis on individualizing HbA1c goals and selecting drugs based on clinical profiles to maximize benefits and minimize harm.
  These patients will also undergo an intensive 3 to 4 months empowerment program where patients within the same group, and therefore sharing similar profiles, will return to the centre monthly to undergo a 2-3 hour activity session led by diabetes nurses, peer supporters and paramedics. Between medical visits, the nurses or HCA will telephone the patients at least once to provide support, help problem-shoot and remind them of their follow-up schedule.
  Arms: EMERALD
Other: Usual Care — Patients randomised to the usual care group will receive their routine care after the initial baseline comprehensive assessment & explanation of the JADE reports. A repeat comprehensive assessment will then be conducted at year 3.
  Arms: Usual Care

SUMMARY:
This is a pilot translational study aiming to compare the effects of a multi-component care program with personalized drug regimen augmented by behavioural therapy with psychological support and peer influence, led by a diabetes specialist team on metabolic control, psychological health and behaviours in difficult-to-treat type 2 diabetic patients versus usual care.

The study hypothesis is to evaluate a novel individualized, multicomponent care program to optimize glycemic control in difficult-to-treat type 2 diabetic patients.

DETAILED DESCRIPTION:
Diabetic patients are at high risk for co-morbidities which are closely related to disease duration and coexisting cardiovascular risk factors and complications. Data has shown that the following 3 groups of diabetic patients are at extremely high risk for future events:

1. Obese type 2 diabetic patients: Weight control is a major therapeutic challenge which often requires cognitive-psychological-behavioral therapy (CBT) in addition to pharmacological and surgical interventions. After long disease duration, often characterized by the presence of complications, many obese diabetic patients need insulin to control glycemia which put them at risk of further weight gain which sets up a vicious cycle.
2. Young type 2 diabetic patients: In both Pima Indian and Caucasian type 2 diabetic patients, young age of onset substantially increased risk of cardiovascular and renal complications, mainly due to long disease duration. Furthermore, these patients often default follow up or are non-compliant due to competing priorities and lack of symptoms. These young patients also have marked phenotypic heterogeneity characterised by insulin insufficiency and/or obesity with strong family history.
3. Diabetic patients with established cardiovascular-renal complications. In a series of analyses, Chinese type 2 diabetic patients with established cardiovascular and kidney disease had 38% event rates including all-cause death and cardiovascular-renal complications including peripheral vascular disease (PVD) over 5 years.

These 3 groups of patients are difficult to treat with many unmet needs requiring complex treatment regimens, intensive counselling and emotional support.

In a series of studies, the investigators have confirmed the marked benefits of using a team approach to deliver structured care with particular emphasis on continuation of care and periodic reminders on clinical outcomes. Preliminary analysis from our peer support program also demonstrated the benefits of utilizing organized and visual information to communicate personalized risks and targets, further augmented by peer support, to improve risk factor control in type 2 diabetic patients.

ELIGIBILITY:
Inclusion Criteria:

* Obese type 2 diabetic patients: body mass index (BMI) >27 kg/m2 and/or waist circumference (WC) >80cm in women and >90cm in men and HbA1c >8% aged 18-70 years
* Young type 2 diabetic patients: age 35-55 years and HbA1c >8%
* Diabetic patients with established cardiovascular-renal complications: HbA1c >8% and known cardiovascular and renal complications with chronic kidney disease (CKD) stage 3-4 (i.e. estimated glomerular filtration rate <60 to >15 ml/min/ per 1.73m2) aged 18-70 years.

Exclusion Criteria:

* Type 1 diabetes
* Active malignant disease (Patients with malignant disease who have been disease-free for at least 5 years are eligible)
* Life expectancy less than 12 months
* Any medical illness or condition as judged by the investigators as ineligible to participate the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2012-05; Primary Completion 2017-07 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Glycemic control as measured by HbA1c compared to baseline | 36 months
  Outcome measures will be assessed in all 600 patients in the both groups at 1 year and 3 year.

SECONDARY OUTCOMES:
Control of BP compared to baseline. | 36 months
  Outcome measures will be assessed in all 600 patients in both groups at 1 year and 3 year.
Control of low density lipoprotein (LDL) cholesterol compared to baseline. | 36 months
  Outcome measures will be assessed in all 600 patients in the both groups at 1 year and 3 year.
Control of BMI and other obesity indices compared to baseline | 36 months
  Outcome measures will be assessed in all 600 patients in the both groups at 1 year and 3 year.

CONTACTS AND LOCATIONS:
Overall Officials: Juliana Chan, MD, Principal Investigator — Asia Diabetes Foundation
Locations (1):
- DMEC Centre, Prince of Wales Hospital, Shatin, Hong Kong